CLINICAL TRIAL: NCT02923635
Title: A Prospective Comparative Study Between Oncoplastic Breast Surgery and Standard Wide Local Excision:Margin Length and Patient Satisfaction
Brief Title: A Prospective Comparative Study Between Oncoplastic Breast Surgery and Standard Wide Local Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Abdel-samii, Lecturer of General surgery, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006379
Record Dates: First submitted 2016-10-02; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Oncoplastic breast surgery; Standard Wide Local Excision
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Wide Local Excision group (Active Comparator): Group A (35 patients) have standard curative conservative breast surgery without integration of plastic techniques .
  Interventions: Procedure: Standard wide local excision.
- Oncoplastic group (Active Comparator): Group B(35 patients) have curative oncoplastic surgery in which plastic techniques integrated with oncological procedures
  Interventions: Procedure: oncoplastic breast surgery.

INTERVENTIONS:
Procedure: Standard wide local excision. — Excision of breast cancer without integration of plastic technique
  Arms: Standard Wide Local Excision group
Procedure: oncoplastic breast surgery. — Integration of plastic techniques with oncological surgery for resection of breast cancer.
  Arms: Oncoplastic group

SUMMARY:
The aim of this study is to asses the oncological safety of oncoplastic breast surgery, and its impact on patient satisfaction.

DETAILED DESCRIPTION:
This non-randomized prospective trial was conducted on70 female patients presented to tertiary breast unit-Ain Shams University hospitals with breast cancer during the period from September 2012 to February 2013. All patients sharing in the study signed an informed consent that was approved in the ethical committee held on April 2012. Patients were classified in two groups each one 35 patients: group (A) standard wide local excision and group (B) oncoplastic group. Standard wide local excision done by general breast surgeons while oncoplastic surgeries done by breast surgeon assisted by plastic surgeon. The following data were recorded: Age, family history, margin length, weight and volume of the specimen, margin status and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with macromastia in oncoplastic group.
* Tumors >20% of breast volume in oncoplastic group.
* Young patients in oncoplastic group
* Tumors in medial or central quadrants in oncoplastic group

Exclusion Criteria:

* Patients >60 years.
* Patients with co-morbidities in oncoplastic group.
* Tumors >20% of breast volume in standard group.
* Tumors in medial or central quadrants in standard group

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Margins in all specimens measured in millimeters | Two years

SECONDARY OUTCOMES:
Patient satisfaction assessed using questionnaire | two years

IPD SHARING:
Plan to Share IPD: Undecided